CLINICAL TRIAL: NCT02937480
Title: Efficacy of Task-specific Training on Physical Activity Levels of People With Stroke: A Randomized Controlled Trial
Brief Title: Efficacy of Task-specific Training on Physical Activity Levels Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Christina Danielli Coelho de Morais Faria, Doctor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 51453915.1.0000.5149
Record Dates: First submitted 2016-09-18; First posted 2016-10-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: stroke; physical activity; task performance; clinical protocol
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Task-specific training
  Interventions: Other: Task-specific training
- Control group (Sham Comparator): Global stretching, memory exercises, health care orientation
  Interventions: Other: Global stretching, memory exercises, health care orientation

INTERVENTIONS:
Other: Task-specific training — The task-specific training will be composed by 30 minutes for upper limb and 30 minutes for lower limb tasks. Subjects will performed five minutes of exercise in each station of the circuit and only the last station will last 10 minutes and will involve a walking training with auditory stimulation. Individuals will be encouraged to work as hard as possible at each station and verbal feedback and instructions aimed at improving performance will be taken. Between each task, the participants will be allowed to rest for at least 1-2 minutes, and individual adjustments will be carried out for better adaptations to the training.
  Other Names: Task-oriented training
  Arms: Experimental group
Other: Global stretching, memory exercises, health care orientation — The control intervention will be composed by 40 minutes for global stretching, 20 minutes of memory exercises and health care orientation
  Arms: Control group

SUMMARY:
The majority of people after stroke demonstrate mobility limitations, which may reduce their physical activity levels. Task-specific training has shown to be an effective intervention to improve mobility in individuals with stroke, however, little is known about the impact of this intervention on levels of physical activity. The main objective will be to investigate the efficacy of a task-specific training, focused on both upper and lower limbs, in improving physical activity levels and mobility in individuals with stroke. The secondary objective will be to investigate the effect of the training, in improving muscle strength, exercise capacity, and quality of life. A randomized controlled trial with blinded assessment will assign eligible participants to either: 1) experimental group or 2) control group. Participants will receive interventions three times per week over 12 weeks. The experimental group will undertake task-specific training, while the control group will undertake global stretching and memory exercises, and health education sessions. Primary outcomes will include measures of physical activity levels and mobility, whereas secondary outcomes will be muscle strength, exercise capacity, and quality of life. The outcomes will be measured at baseline, 12 weeks post-intervention, and four and 12 weeks follow-up. The findings of this trial have the potential to provide important insights regarding the effects of task-specific training, focused on both upper and lower limbs, in preventing secondary post-stroke complications and improving the participants' general health through changes in physical activity levels.

DETAILED DESCRIPTION:
The sample size was calculated to detect a between-group difference of 0.15 m/s in gait speed, with 80% power, at a two-tailed significance level of 0.05. In an RCT with a similar population and intervention (Yang et al. 2006) gait speed for the control and experimental groups at baseline was 0.78±0.14 m/s and 0.84±0.13 m/s and after were 0.78±0.15 m/s (p=0.8) and 0.93±0.14 m/s (p<.001), respectively. Based on these values, 15 participants per group will be required (a total of 30 participants). Assuming a dropout rate of 15%,66 a total of 36 participants will be recruited (18 per group).

Data analyses will be performed by the SPSS for Windows® (release 17.0, SPSS Inc., Chicago, IL, USA). Descriptive statistics will be carried-out for all outcome variables. Differences between the groups at baseline will be investigated with the independent Student's t-tests for all variables related to the demographic and clinical characteristics. If differences between the groups at baseline exist, analysis of covariance will be used to eliminate the influence of extraneous factors.

The effects of the interventions will be analysed in two ways, namely from the data collected and by intention-to-treat analyses, where the last available value in the dropouts will be carried forward to represent the missing data. Analyses of variance with repeated measures (2×4) will be employed to investigate the mean and interaction effects between the groups (intervention×control) and the time (preintervention, postintervention, and follow-up) for the primary and secondary outcomes. Group descriptions will be presented as mean (SD) and effect sizes with 95% confidence intervals (CIs) will be reported.

The effect sizes will be calculated to determine the magnitude of the differences between the groups. The differences between the two mean values will be expressed in units of their SD, expressed as Cohen's d, or mean results for the experimental group minus the mean results for the control group, divided by the SD of the control group. Effect sizes between 0.2 and 0.5 will be considered small; between 0.5 and 0.8, medium; and above 0.8, large.

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of first or recurrent stroke more than six months since the onset of their strokes;
* are older than 19 years of age;
* are able to independently walk 10 m with or without walking aid devices;
* have tone of elbow flexor muscles below 4 on modified Ashworth scale;
* are inactive or insufficient, based on Centers for Disease Control and Prevention criteria;
* get medical permission for physical activity practice

Exclusion Criteria:

* have severe cognitive deficits, as assessed by the mini-mental state exam and/or language problems (comprehensive afasia), as evaluated by simple motor commands ("lift your nonparetic upper limb and open your hand"), which might prevent them from following instructions during the data collection and/or the interventions;
* have history of severe heart disease and/or uncontrolled blood pressure;
* have pain and/or other adverse health conditions which might affect the performance in the intervention program, such as vestibular disturbances, severe arthritis, or other neurological disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Physical activity levels - physical activity monitor | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Physical activity levels will be assessed by a physical activity monitor (SenseWear®, BodyMedia, Pittsburgh, USA).
Change from baseline in Physical activity levels - Human Activity Profile | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Physical activity levels will be assessed by Human Activity Profile.
Change from baseline in Mobility - Gait speed | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Mobility will be assessed by gait speed.
Change from baseline in Mobility - TEMPA | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Mobility will be assessed by TEMPA test.

SECONDARY OUTCOMES:
Change from baseline in Muscle strength | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Muscle strength will be assessed by hydraulic handgrip dynamometer SAEHAN® (SAEHAN Corporation, Korea, Model SH5001) and digital handheld dynamometer Microfet2® (Hoggan Health Industries, UT, USA).
Change from baseline in Exercise capacity | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Exercise capacity will be assessed by six minute walk test.
Change from baseline in Quality of life | At baseline, after 12 weeks post-intervention, four and 12 weeks of follow-up
  Quality of life will be assessed by Stroke specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Danielli CM Faria, Doctor, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendis S. Stroke disability and rehabilitation of stroke: World Health Organization perspective. Int J Stroke. 2013 Jan;8(1):3-4. doi: 10.1111/j.1747-4949.2012.00969.x. No abstract available. PMID 23280261
- [Background] Ovbiagele B, Goldstein LB, Higashida RT, Howard VJ, Johnston SC, Khavjou OA, Lackland DT, Lichtman JH, Mohl S, Sacco RL, Saver JL, Trogdon JG; American Heart Association Advocacy Coordinating Committee and Stroke Council. Forecasting the future of stroke in the United States: a policy statement from the American Heart Association and American Stroke Association. Stroke. 2013 Aug;44(8):2361-75. doi: 10.1161/STR.0b013e31829734f2. Epub 2013 May 22. PMID 23697546
- [Background] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Martins SC, Pontes-Neto OM, Alves CV, de Freitas GR, Filho JO, Tosta ED, Cabral NL; Brazilian Stroke Network. Past, present, and future of stroke in middle-income countries: the Brazilian experience. Int J Stroke. 2013 Oct;8 Suppl A100:106-11. doi: 10.1111/ijs.12062. Epub 2013 May 22. PMID 23692595
- [Background] Morris JH, Macgillivray S, McFarlane S. Interventions to promote long-term participation in physical activity after stroke: a systematic review of the literature. Arch Phys Med Rehabil. 2014 May;95(5):956-67. doi: 10.1016/j.apmr.2013.12.016. Epub 2014 Jan 1. PMID 24389402
- [Background] Fini NA, Holland AE, Keating J, Simek J, Bernhardt J. How is physical activity monitored in people following stroke? Disabil Rehabil. 2015;37(19):1717-31. doi: 10.3109/09638288.2014.978508. Epub 2014 Nov 6. PMID 25374044
- [Background] Resnick B, Michael K, Shaughnessy M, Nahm ES, Kobunek S, Sorkin J, Orwig D, Goldberg A, Macko RF. Inflated perceptions of physical activity after stroke: pairing self-report with physiologic measures. J Phys Act Health. 2008 Mar;5(2):308-18. doi: 10.1123/jpah.5.2.308. PMID 18382039
- [Background] Caspersen CJ, Powell KE, Christenson GM. Physical activity, exercise, and physical fitness: definitions and distinctions for health-related research. Public Health Rep. 1985 Mar-Apr;100(2):126-31. PMID 3920711
- [Background] Strath SJ, Kaminsky LA, Ainsworth BE, Ekelund U, Freedson PS, Gary RA, Richardson CR, Smith DT, Swartz AM; American Heart Association Physical Activity Committee of the Council on Lifestyle and Cardiometabolic Health and Cardiovascular, Exercise, Cardiac Rehabilitation and Prevention Committee of the Council on Clinical Cardiology, and Council. Guide to the assessment of physical activity: Clinical and research applications: a scientific statement from the American Heart Association. Circulation. 2013 Nov 12;128(20):2259-79. doi: 10.1161/01.cir.0000435708.67487.da. Epub 2013 Oct 14. PMID 24126387
- [Background] Warren JM, Ekelund U, Besson H, Mezzani A, Geladas N, Vanhees L; Experts Panel. Assessment of physical activity - a review of methodologies with reference to epidemiological research: a report of the exercise physiology section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2010 Apr;17(2):127-39. doi: 10.1097/HJR.0b013e32832ed875. PMID 20215971
- [Background] Pollock A, Baer G, Campbell P, Choo PL, Forster A, Morris J, Pomeroy VM, Langhorne P. Physical rehabilitation approaches for the recovery of function and mobility following stroke. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD001920. doi: 10.1002/14651858.CD001920.pub3. PMID 24756870
- [Background] Chae J, Johnston M, Kim H, Zorowitz R. Admission motor impairment as a predictor of physical disability after stroke rehabilitation. Am J Phys Med Rehabil. 1995 May-Jun;74(3):218-23. doi: 10.1097/00002060-199505000-00007. PMID 7779333
- [Background] Ashe MC, Miller WC, Eng JJ, Noreau L; Physical Activity and Chronic Conditions Research Team. Older adults, chronic disease and leisure-time physical activity. Gerontology. 2009;55(1):64-72. doi: 10.1159/000141518. Epub 2008 Jun 20. PMID 18566534
- [Background] English C, Hillier SL. Circuit class therapy for improving mobility after stroke. Cochrane Database Syst Rev. 2010 Jul 7;2010(7):CD007513. doi: 10.1002/14651858.CD007513.pub2. PMID 20614460
- [Background] Tiedemann A, Sherrington C, Dean CM, Rissel C, Lord SR, Kirkham C, O'Rourke SD. Predictors of adherence to a structured exercise program and physical activity participation in community dwellers after stroke. Stroke Res Treat. 2012;2012:136525. doi: 10.1155/2012/136525. Epub 2011 Oct 11. PMID 22007351
- [Background] Alzahrani MA, Dean CM, Ada L. Ability to negotiate stairs predicts free-living physical activity in community-dwelling people with stroke: an observational study. Aust J Physiother. 2009;55(4):277-81. doi: 10.1016/s0004-9514(09)70008-x. PMID 19929771
- [Background] French B, Thomas L, Leathley M, Sutton C, McAdam J, Forster A, Langhorne P, Price C, Walker A, Watkins C. Does repetitive task training improve functional activity after stroke? A Cochrane systematic review and meta-analysis. J Rehabil Med. 2010 Jan;42(1):9-14. doi: 10.2340/16501977-0473. PMID 20111838
- [Background] Jeon BJ, Kim WH, Park EY. Effect of task-oriented training for people with stroke: a meta-analysis focused on repetitive or circuit training. Top Stroke Rehabil. 2015 Feb;22(1):34-43. doi: 10.1179/1074935714Z.0000000035. Epub 2015 Jan 21. PMID 25776119
- [Background] Rensink M, Schuurmans M, Lindeman E, Hafsteinsdottir T. Task-oriented training in rehabilitation after stroke: systematic review. J Adv Nurs. 2009 Apr;65(4):737-54. doi: 10.1111/j.1365-2648.2008.04925.x. Epub 2009 Feb 9. PMID 19228241
- [Background] Mudge S, Barber PA, Stott NS. Circuit-based rehabilitation improves gait endurance but not usual walking activity in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Dec;90(12):1989-96. doi: 10.1016/j.apmr.2009.07.015. PMID 19969159
- [Background] Dean CM, Rissel C, Sherrington C, Sharkey M, Cumming RG, Lord SR, Barker RN, Kirkham C, O'Rourke S. Exercise to enhance mobility and prevent falls after stroke: the community stroke club randomized trial. Neurorehabil Neural Repair. 2012 Nov-Dec;26(9):1046-57. doi: 10.1177/1545968312441711. Epub 2012 Apr 27. PMID 22544817
- [Background] Michael K, Goldberg AP, Treuth MS, Beans J, Normandt P, Macko RF. Progressive adaptive physical activity in stroke improves balance, gait, and fitness: preliminary results. Top Stroke Rehabil. 2009 Mar-Apr;16(2):133-9. doi: 10.1310/tsr1602-133. PMID 19581199
- [Background] Pang MY, Eng JJ, Dawson AS, McKay HA, Harris JE. A community-based fitness and mobility exercise program for older adults with chronic stroke: a randomized, controlled trial. J Am Geriatr Soc. 2005 Oct;53(10):1667-74. doi: 10.1111/j.1532-5415.2005.53521.x. PMID 16181164
- [Background] Ainsworth B, Cahalin L, Buman M, Ross R. The current state of physical activity assessment tools. Prog Cardiovasc Dis. 2015 Jan-Feb;57(4):387-95. doi: 10.1016/j.pcad.2014.10.005. Epub 2014 Oct 31. PMID 25446555
- [Background] Manns PJ, Dunstan DW, Owen N, Healy GN. Addressing the nonexercise part of the activity continuum: a more realistic and achievable approach to activity programming for adults with mobility disability? Phys Ther. 2012 Apr;92(4):614-25. doi: 10.2522/ptj.20110284. Epub 2011 Dec 9. PMID 22156025
- [Background] English C, Manns PJ, Tucak C, Bernhardt J. Physical activity and sedentary behaviors in people with stroke living in the community: a systematic review. Phys Ther. 2014 Feb;94(2):185-96. doi: 10.2522/ptj.20130175. Epub 2013 Sep 12. PMID 24029302
- [Background] Pang MY, Harris JE, Eng JJ. A community-based upper-extremity group exercise program improves motor function and performance of functional activities in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2006 Jan;87(1):1-9. doi: 10.1016/j.apmr.2005.08.113. PMID 16401430